CLINICAL TRIAL: NCT07351552
Title: The Effect of Frailty in Geriatric Patients on Hypotension Observed After Anesthesia Induction
Brief Title: The Effect of Frailty on Hypotension After Anesthesia Induction
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, EMİNE ASLANLAR, associated professor, Selcuk University
Other Study IDs: frailty, anesthesia induction
Record Dates: First submitted 2025-12-17; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Fraility; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is defined as a state of weakness resulting from a decrease in physiological reserves due to physiological changes, diseases, and/or malnutrition associated with advancing age. Frail older adults face increased mortality, morbidity, and healthcare costs when exposed to stressors, making this issue increasingly important. The FRAIL Scale, developed by Morley et al. , is a 5-item measure that assesses frailty. The FRAIL Scale has been validated in many countries and has been proven to be an effective method for detecting frailty. This scale assesses the patient's fatigue, resistance, mobility, weight loss, and other diseases. In the 5-item FRAIL scale, patients receive 0 or 1 point based on their answers, and a total of 0 points is considered non-frail, 1-2 points is considered pre-frail, and >2 points is considered frail.

Frailty is associated with a higher risk of postoperative complications. Rothenberg and colleagues reported in a study involving more than 400,000 patients that frailty doubles the risk of postoperative complications .

Hypotension following anesthesia induction is a common complication in geriatric patients. Decreased cardiopulmonary reserve with age leads to an exaggerated drop in blood pressure during induction .

In this study, the investigators aimed to determine the effect of frailty level in geriatric patients on hypotension observed after anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who do not have difficulty communicating,
* have good cognitive function,
* scheduled for surgery under general anesthesia

Exclusion Criteria:

* Patients admitted for surgery in emergency situations
* Patients with active malignancy
* Patients with physical disabilities and impairments (limb amputations, stroke sequelae, unable to speak, hearing problems)
* Patients with acute infections
* Patients with acute illnesses (decompensated congestive heart failure, recent myocardial infarction/stroke, COPD exacerbation)
* Patients who have been hospitalized or undergone surgery within the last month
* Patients with advanced dementia
* Patients who are unable to provide a medical history or cooperate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over the age of 65 undergoing elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The effect of fragility level on hypotension observed after anesthesia induction | 20 minutes

IPD SHARING:
Plan to Share IPD: Undecided